CLINICAL TRIAL: NCT04768218
Title: Blue Light Imaging System for the Diagnosis of Precancerous Conditions: European Multicenter Validation Study
Brief Title: BLI for the Diagnosis of Precancerous Conditions
Status: Completed | Type: Observational
Sponsor: Instituto Portugues de Oncologia, Francisco Gentil, Porto (Other)
Responsible Party: Sponsor
Other Study IDs: 207/020
Record Dates: First submitted 2021-02-17; First posted 2021-02-24 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2023-12

CONDITIONS: Gastric Cancer; Preneoplastic Condition; Early Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms; Precancerous Conditions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Introduction: Traditionally, White Light Endoscopy (WLE), enhanced by biopsies following the updated Sydney system guidelines, has been the benchmark for diagnosing and classifying gastric preneoplastic conditions. Nevertheless, the pronounced interobserver variability and the often weak correlation between endoscopic observations and histopathological results have driven the increasing adoption of virtual chromoendoscopy (VCE). VCE technologies have demonstrated greater effectiveness in identifying these conditions compared to WLE, with Narrow Band Imaging (NBI) being particularly notable. Significantly, NBI has played a key role in validating the Endoscopic Grading of Gastric Intestinal Metaplasia (EGGIM) system. However, data on the effectiveness of other VCE technologies in this domain is relatively sparse in Europe, specifically with Blue Light Imaging (BLI), despite the promising diagnostic performance demonstrated with this technology.

Primary aim: to assess the diagnostic accuracy of BLI and to externally validate the applicability of EGGIM classification for staging GIM.

Material and methods: a multicentric cohort study will be performed involving centres from two European countries (Portugal, Italy). Consecutive patients performing upper gastrointestinal endoscopy will be evaluated by WLE and BLI. Random biopsies or targeted plus random biopsies will be performed in order to determine de accuracy of BLI system to detect and stage GIM.

Expected results: We anticipate that BLI would enable us to assess the extension of GIM without the need for biopsies. If observed, this would overall improve the upper GI endoscopy accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Individuals older than 18 years.
* Indication to submit diagnostic or surveillance upper GI endoscopy.

Exclusion Criteria:

* History of previous gastric surgery.
* History of previous gastric cancer.
* Contraindications to biopsies.
* Individuals unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients referred to the endoscopy department of a tertiary care center for screening or surveillance upper gastrointestinal endoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
To determine the inter-observer agreement and accuracy of BLI system for the diagnosis and endoscopic staging of GIM | During the 3 months after finishing histopathological analysis of biopsies (an average of 17 months)
  For accuracy: A per-biopsy analysis will be performed comparing diagnostic perception per site biopsied (ie, accuracy of WLE or BLI for each site observed vs that result).
  For inter-observer agreement: after following educational set, inter-observer agreement for WLE and BLI will be assessed (see phase 2).
To externally validate the EGGIM score classification using BLI | During the 12 months after finishing histopathological analysis of biopsies (an average of 17 months)
  For accuracy: A per-patient analysis will be performed comparing WLE and BLI accuracy for Operative Link on Gastritis Assessment for Intestinal Metaplasia (OLGIM) III/IV (ie, accuracy of EGGIM estimated by each endoscopist using WLE or BLI towards OLGIM III/IV).
  For inter-observer agreement: after completion phase 3, video records will be assessed by 1 endoscopist and inter-observer agreement for EGGIM classification, using BLI system, will be evaluated

CONTACTS AND LOCATIONS:
Locations (1):
- Marta Rodriguez, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No